CLINICAL TRIAL: NCT07005076
Title: Investigation of the Effects of Technology-Assisted Exercises in Individuals With Chronic Neck Pain
Brief Title: Tech-Assisted Exercise Training in Chronic Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Fatma Eken, Research asistant, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-481633
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Chronic Neck Pain; Exercise Training Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The treatment process for the control group consisted of hot therapy and TENS application before the exercises, followed by an exercise program including neck range of motion exercises, neck strengthening exercises, stretching exercises, scapular retraction, etc.
- Experimental Group (Experimental): The program will be implemented over four weeks, three days a week, with a duration of 40-45 minutes per day. In addition to conventional treatment, an exercise program prepared with a light reaction time measurement and exercise set will be implemented.
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — Participants in the experimental group will participate in a conventional exercise program similar to the control group, but with the addition of a technology-assisted exercise program. The intervention group will receive training with a reaction time measurement set using lights and an exercise set. The reaction time measurement and exercise set will be used, where light pods are placed in different positions, such as on a table, mirror, and floor, and patients will be instructed to extinguish the lit light as quickly as possible. The difficulty level of the sessions will be progressively increased by adjusting factors such as the duration of light activation, colors, the number of illuminated pods, their placement locations, and the distance between them.
  Other Names: Tech-Assisted Training
  Arms: Experimental Group

SUMMARY:
In this study, women with chronic neck pain residing in Afyonkarahisar, Turkey, will participate in an exercise-based intervention. Both the control and experimental groups will engage in conventional exercise programs; however, the experimental group will also receive an additional technology-assisted exercise program. It is anticipated that these interventions will positively impact participants' daily living activities and functional abilities. The study aims to assess whether the inclusion of technology-supported exercises leads to superior outcomes compared to conventional exercises alone. The findings are expected to provide valuable evidence on the effectiveness of integrating technology-assisted exercise programs into physiotherapy and rehabilitation practices for women with chronic neck pain.

DETAILED DESCRIPTION:
Considering the complex nature of chronic pain, it is believed that integrating exercise approaches with technology may enhance the effectiveness of exercise programs, increase participation and its sustainability, support the continuity of overall health and functional outcomes, and have positive effects on behavior change. The light-based exercise set for measuring reaction time is frequently preferred in clinical settings. The device uses small, illuminated pods controlled by an application, providing visual cues that promote both physical and cognitive activity. The individual aims to deactivate the lit pods as quickly as possible. Due to its interactive and enjoyable nature, it is commonly used across a wide range of populations-from pediatric to geriatric-especially among athletes. Technology-focused approaches, compared to traditional exercise practices, are believed to positively influence patients' active participation in the treatment process through a more innovative and engaging experience.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific neck pain diagnosis
* Having neck pain persisting for at least 3 months
* Having the ability to speak and comprehend Turkish fluently
* A pain score of 3 or higher according to the Numerical Rating Scale
* A score of 5 or higher on the Neck Disability Index

Exclusion Criteria:

* Having a history of spinal surgery.
* Having an additional musculoskeletal disorder affecting the cervical region and upper extremities (e.g., scoliosis, rheumatoid arthritis, fibromyalgia, etc.).
* Receiving physical therapy and/or other treatments for any reason within the last 6 months.
* Having a diagnosed psychiatric disorder.
* Having a vestibular pathology.
* Having visual problems despite using visual aids.
* Being pregnant.
* Having a neurological deficit that may affect balance.
* Discontinuing or being unable to complete the treatment process.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | From enrollment to the end of treatment at 4 weeks
  Patients will be asked to mark the number between 0 and 10 that best corresponds to the intensity of their pain.
G-Walk Wireless Movement Analysis System | From enrollment to the end of treatment at 4 weeks
  G-Walk is a wireless system used to assess gait, balance, and functional mobility through motion sensors placed on the lower back. While wearing the G-Walk device, the participant walks at a normal pace between two markers placed 10 meters apart. Furthermore, static balance will be assessed by having the participant maintain a one-legged stance for 30 seconds.
Modified Four Square Step Test | From enrollment to the end of treatment at 4 weeks
  The Modified Four Square Step Test (mFSST) is used to assess dynamic balance and the ability to step in multiple directions. During the test procedure, four strips, each measuring 90 cm in length, are arranged on the floor to form a square, with each quadrant labeled from 1 to 4. The participant is instructed to step through each quadrant first in a clockwise direction and then in a counterclockwise direction, ensuring continuous forward gaze and avoiding contact with the strips throughout the test.

CONTACTS AND LOCATIONS:
Overall Officials: FATMA EKEN, Principal Investigator — Afyonkarahisar Sağlık Bİlimleri Üniversitesi
Locations (1):
- Afyonkarahisar Health Sciences University, Merkez, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No